CLINICAL TRIAL: NCT00111826
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of Efficacy and Safety of the Celacade™ System in Improving Walking Distance in Patients With Intermittent Claudication Secondary to Peripheral Arterial Disease
Brief Title: SIMPADICO - Study of Immune Modulation Therapy in Peripheral Arterial Disease and Intermittent Claudication Outcomes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Vasogen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0101
Record Dates: First submitted 2005-05-25; First posted 2005-05-26 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2007-11

CONDITIONS: Peripheral Arterial Disease; Arterial Occlusive Diseases; Intermittent Claudication
Keywords: Intermittent Claudication; Peripheral Arterial Disease; Immune modulation therapy; Inflammation
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases; Intermittent Claudication; Inflammation

INTERVENTIONS:
Device: Celacade™ system

SUMMARY:
The purpose of this study is to assess the effects of the Celacade™ system in patients with intermittent claudication.

DETAILED DESCRIPTION:
SIMPADICO was a multicenter, randomized, double-blind, placebo-controlled trial that enrolled 553 patients with claudication at 50 sites in Canada and the United States. The mean (±SD) patient age was 67±10 years; 72% were males. The duration of claudication was 6.0±6.1 years at entry; 91% had a history of smoking and 34% were current smokers; 36.5% had diabetes. Resting ABI was 0.59+0.14; baseline ICD was 132±104 and ACD 307±209 meters. Results showed that there was no increase in ACD or ICD at 26 weeks with immune modulation therapy (IMT using the Celacade™ system, Vasogen Inc.) compared to placebo and no measurable improvement in quality of life with IMT compared to placebo. However, there was a significant decrease in CRP (high sensitivity assay) in) in the IMT group compared to the placebo group. Conclusion: Immune modulation therapy did not improve walking distance in patients with symptomatic peripheral arterial disease but the decrease in CRP suggests a biologic effect of IMT and will warrant further study.

Reference: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Immune Modulation Therapy in Patients with Symptomatic Peripheral Arterial Disease: The SIMPADICO Trial. Author: Jeffrey W. Olin, Mount Sinai School of Medicine, New York, NY. Presented at Smaller Trial Late-Breaking Clinical trials I, Sunday March 12, 2006. American College of Cardiology 55th Annual Scientific Sessions, March 11-14, 2006, Atlanta, GA.

ELIGIBILITY:
Inclusion Criteria:

* History of intermittent claudication (Fontaine stage II) due to peripheral arterial disease, which has been stable (both clinically and therapeutically) for 3 months prior to screening.
* Resting ankle-brachial index (ABI) in at least one limb ≤ 0.85. For diabetics with falsely elevated ABI due to non-compressible tibial arteries, the toe brachial index (TBI) will be measured and has to be ≤ 0.7 at rest.
* An absolute claudication distance (ACD) of≥ 50 meters confirmed on two consecutive visits at least one week apart. The change in ACD between the two consecutive assessments (i.e. Visit 0 and 1 or Visit 1 and 2) has to be within ± 20%.
* Walking distance must be limited by IC, which will be confirmed by a ≥ 20% decrease in ABI in the worse claudicating limb immediately following the screening treadmill tests. The worse claudicating limb (or "index leg") will be defined either as (1) the most symptomatic leg or (2) the leg with the lowest resting ABI and documented prior to the first (pre-screening) treadmill test. Post-exercise and resting ABIs will be compared within the same leg at each screening treadmill test. This criterion will not apply to diabetics with non-compressible tibial arteries (i.e. only the resting TBI will be measured in these patients).
* Age ≥40 years

Exclusion Criteria:

* Women who are pregnant, lactating, or of childbearing potential not using accepted contraceptive methods, as assessed by the investigator.
* Clinically relevant abnormal findings in the clinical history or physical examination at the screening assessment that would interfere with the objectives of the study or that would, in the investigator's opinion, preclude safe completion of the study. Abnormal findings could include: hepatitis, HIV infection, AIDS, other immune deficiency syndromes, serious active infections, gastrointestinal tract bleeding or any severe or acute concomitant illness or injury.
* Critical limb ischemia (CLI) defined as ischemic rest pain, ulcerative lesions or gangrene [Rutherford-Becker Classification Grade II-III (corresponding to Fontaine stage III-IV)].
* Previous endovascular or surgical revascularization within 6 months prior to study entry or anticipated during the first 6 months of the study.
* Active inflammatory vascular disease (e.g. Buerger's disease).
* Major peripheral neuropathies, including severe diabetic neuropathy to the extent that it may interfere with the evaluation of claudication.
* Any condition that limits walking ability, other than claudication (e.g. arthritis, angina, chronic obstructive pulmonary disease [COPD], etc.)
* Malignancy within five years prior to screening. Basal cell carcinoma, provided that it is neither infiltrating nor sclerosing, and carcinoma in situ of the cervix are exemptions.
* Organ transplant recipients.
* Allergy to sodium citrate, or any "caine" type of local anesthetic.
* Systemic corticosteroids, antineoplastics and immunosuppressive drug therapy (e.g. cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.), DNA depleting or cytotoxic drugs taken within 4 weeks prior to study treatment.
* Currently taking medications indicated for intermittent claudication (i.e. pentoxifylline or cilostazol). To be eligible, patient must not have taken these medications for at least 8 weeks prior to study enrollment.
* Participation in another study involving an investigational or licensed drug or device in the 4 weeks preceding enrollment or during this study.
* Previous Celacade™ treatment.
* Any other medical, social, or geographical factor, which would make it unlikely that the patient will comply with study procedures (e.g. alcohol abuse, lack of permanent residence, severe depression, disorientation, distant location, and a history of non-compliance).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2003-01; Study Completion 2005-12

PRIMARY OUTCOMES:
Absolute claudication distance (ACD)

SECONDARY OUTCOMES:
Health-related quality of life
Functional status
Combined incidence of peripheral arterial disease (PAD)-related clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Shannon, MD, Study Director — Vasogen Inc.